CLINICAL TRIAL: NCT02416791
Title: Robotic Therapy and Transcranial Direct Current Stimulation in Patients With Stroke
Acronym: ROTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of low recruitment rates
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 513.207
Record Dates: First submitted 2015-02-20; First posted 2015-04-15 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2015-12

CONDITIONS: Stroke
Keywords: robotic therapy; transcranial direct current stimulation
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active tDCS + robotic therapy + physical therapy (Active Comparator): Active tDCS (transcranial direct current stimulation) will be applied prior to the robotic training. After robot training, the patient will receive physical therapy for 40 minutes.
  Number of treatment sessions: 18 (3 times a week, for 6 weeks).
  Interventions: Device: Robotic Therapy; Device: Active tDCS; Other: Physical Therapy
- sham tDCS + robotic therapy + physical therapy (Active Comparator): Sham tDCS (transcranial direct current stimulation) will be applied prior to robotic training. After robot training, the patient will receive physical therapy for 40 minutes.
  Number of treatment sessions: 18 (3 times a week, for 6 weeks).
  Interventions: Device: Robotic Therapy; Device: Sham tDCS; Other: Physical Therapy
- sham tDCS + physical therapy + occupational therapy (Experimental): Sham tDCS (transcranial direct current stimulation) will be applied prior to conventional therapy (40 minutes of physical therapy and 40 minutes of occupational therapy) Number of treatment sessions: 18 (3 times a week, for 6 weeks).
  Interventions: Device: Sham tDCS; Other: Physical Therapy; Other: Occupational Therapy

INTERVENTIONS:
Device: Robotic Therapy — Robotic therapy (MIT - Manus, Interactive Motion Technologies) will be administered for 40 minutes to the paretic upper limb.
  Arms: Active tDCS + robotic therapy + physical therapy; sham tDCS + robotic therapy + physical therapy
Device: Active tDCS — Active tDCS will be applied with the cathode positioned over the ipsilesional primary motor cortex and the anode over the contralateral supraorbital region for 20 minutes (1mA).
  Arms: Active tDCS + robotic therapy + physical therapy
Device: Sham tDCS — In sham tDCS, no current will be delivered through the tDCS device.
  Arms: sham tDCS + physical therapy + occupational therapy; sham tDCS + robotic therapy + physical therapy
Other: Physical Therapy — Physical therapy will be administered for 40 minutes.
Other: Occupational Therapy — Occupational therapy will be administered for 40 minutes.
  Arms: sham tDCS + physical therapy + occupational therapy

SUMMARY:
Stroke is the second cause of death worldwide and represented the first cause of death in Brazil between 2006 and 2010. Most patients survive, and there is a need to develop cost-effective rehabilitation strategies to decrease the burden of disability from stroke. This study addresses this important issue, by combining two different interventions in the early phase post-stroke: robotic therapy associated or not with transcranial direct current stimulation (tDCS), as adjuvant interventions to conventional physical therapy, for motor upper limb rehabilitation.

DETAILED DESCRIPTION:
Our main goal is to confirm the safety of robotic therapy associated with active tDCS and conventional therapy, compared to robotic therapy associated with sham tDCS and to conventional therapy, and to conventional therapy alone, for upper limb rehabilitation in an early phase (3-9 weeks) after stroke. Patients will be randomized to receive one of these three treatments, 3 times per week, for 6 weeks.

Data about eventual adverse effect will be collected in each session of treatment. The working hypothesis is that robotic therapy associated with active tDCS and conventional therapy will be as safe as robotic therapy associated with conventional therapy, and as conventional therapy alone.

We will aso preliminarily evaluate the efficacy of robotic therapy associated with active tDCS and conventional therapy, compared to robotic therapy associated with sham tDCS and to conventional therapy alone, in improvement of upper limb motor impairment.

Our secondary goals are: 1) To evaluate safety and upper limb motor impairments in patients submitted to each of the three interventions, 6 months after end of treatment; 2) To compare effects of the abovementioned interventions on disability, spasticity and quality of life, in patients at an early stage after stroke, immediately after treatment and 6 months later.

The working hypothesis is that the association of robotic therapy, tDCS and conventional therapy will lead to better outcomes than robotic therapy and conventional therapy, or conventional therapy alone.

Patients will be assessed before the first session and after the last session of treatment, as well as 6 months after the last session of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke onset 3 - 9 weeks before the recruiting, confirmed by computed tomography or magnetic resonance imaging.
* Moderate to severe motor impairment of an upper limb, defined as a score between 7 - 42 on the Upper Limb Subscale of Fugl Meyer Assessment of Sensorimotor Recovery after stroke.
* Ability to provide written informed consent (patient ou legal representative)
* Ability to comply with the schedule of interventions and evaluations in the protocol.

Exclusion Criteria:

* Severe spasticity at the paretic elbow, wrist or fingers, defined as a score of > 3 on the Modified Ashworth Spasticity Scale.
* Upper limb plegia
* Uncontrolled medical problems such as end-stage cancer or renal disease
* Pregnancy
* Seizures, except for a single seizure during the first week post stroke
* Pacemakers
* Other neurological disorders such as Parkinson's disease
* Psychiatric illness including severe depression
* Aphasia ou severe cognitive deficits that compromise comprehension of the experimental protocol or ability to provide consent.
* Hemineglect
* Drugs that interfere on cortical excitability, except for antidepressants
* Cerebellar lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana B Conforto, MD Phd, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS + Robotic Therapy + Physical Therapy: Active tDCS (transcranial direct current stimulation) will be applied prior to the robotic training. After robot training, the patient will receive physical therapy for 40 minutes.
  Number of treatment sessions: 18 (3 times a week, for 6 weeks).
  Robotic Therapy: Robotic therapy (MIT - Manus, Interactive Motion Technologies) will be administered for 40 minutes to the paretic upper limb.
  Active tDCS: Active tDCS will be applied with the cathode positioned over the ipsilesional primary motor cortex and the anode over the contralateral supraorbital region for 20 minutes (1mA).
  Physical Therapy: Physical therapy will be administered for 40 minutes.
- Sham tDCS + Robotic Therapy + Physical Therapy: Sham tDCS (transcranial direct current stimulation) will be applied prior to robotic training. After robot training, the patient will receive physical therapy for 40 minutes.
  Number of treatment sessions: 18 (3 times a week, for 6 weeks).
  Robotic Therapy: Robotic therapy (MIT - Manus, Interactive Motion Technologies) will be administered for 40 minutes to the paretic upper limb.
  Sham tDCS: In sham tDCS, no current will be delivered through the tDCS device.
  Physical Therapy: Physical therapy will be administered for 40 minutes.
Period: 6 Weeks
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: 6 Months
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Started | 3 | 3 | 3
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 7
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (15.2) | 53.33 (4.02) | 54.0 (8.52) | 54.22 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 2 | 3 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Back | 2 | 2 | 3 | 7
  Ethnicity: White | 1 | 1 | 0 | 2
  Ethnicity: Asian | 0 | 0 | 0 | 0
Time since stroke [Mean (Standard Deviation); unit: days] | 49.3 (11.1) | 40.0 (16.75) | 36.66 (11.11) | 41.56 (15.21)
Manual dominance [Count of Participants; unit: Participants]
  Right | 3 | 2 | 3 | 8
  Left | 0 | 1 | 0 | 1
Hemisphere lesioned [Count of Participants; unit: Participants]
  Right hemisphere | 0 | 1 | 1 | 2
  Left hemisphere | 3 | 2 | 2 | 7
Upper Extremity Fugl Meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — Motor function subscale was assessed. Scores range from 0 - 66. Lower scores indicate greater severity.
  units on a scale | 19.3 (9.8) | 17.7 (4.2) | 21.7 (7.8) | 18.89 (6.27)
Mini Mental State Exam [Median (Full Range); unit: units on a scale] — Scores range from 0 to 30. Lower scores indicate greater severity.
  units on a scale | 20 [14 to 28] | 27 [23 to 28] | 25 [22 to 29] | 25 [14 to 29]
National Institutes of Health Stroke Scale [Median (Full Range); unit: units on a scale] — Scores range from 0 -42. Higher scores indicate greater severity.
  units on a scale | 6 [4 to 11] | 6 [2 to 8] | 3 [2 to 4] | 4 [2 to 11]
Modified Rankin Scale [Median (Full Range); unit: units on a scale] — Scores range from 0 to 6. Higher scores indicate greater severity.
  units on a scale | 3 [3 to 4] | 3 [3 to 4] | 3 [3 to 3] | 3 [3 to 4]
Hospital Anxiety and Depression Scale [Median (Full Range); unit: units on a scale] — Both subscales (Anxiety and Depression subscales) were assessed. Scores range from 0 to 42. Higher scores indicate greater severity.
  units on a scale | 8 [7 to 13] | 6 [2 to 9] | 8 [6 to 15] | 8 [2 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Fugl Meyer Assessment
Description: Change in Motor function subscale was assessed. Scores range from 0 to 66. Lower scores indicate greater severity.
Time Frame: 6 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 10.6 (7.3) | 12.3 (11.4) | 22.3 (12.4)

2. Primary Outcome: Percentage of Sessions With Adverse Events
Time Frame: Post treatment (6 weeks from baseline).
Population: RT: robotic therapy; OT: occupational therapy; PT: physical therapy Sham tDCS +RT + PT: 3 participants;each participant was supposed to participate in 18 sessions = 54 sessions in total; there was seven absences and the total number of sessions was 47 for the three patients.
Measure: Number; unit: percentage of sessions
Units Other Than Participants: Number of sessions
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
Number analyzed (Number of sessions) | 53 | 47 | 53
percentage of sessions
  Pain reported during tDCS | 0 | 0 | 1.9
  Fatigue reported during tDCS | 0 | 0 | 0
  Tingling reported during tDCS | 100 | 27.7 | 37.7
  Burning reported during tDCS | 0 | 2.1 | 5.7
  Hot reported during tDCS | 0 | 0 | 0
  Pinching reported during tDCS | 9.4 | 31.9 | 30.2
  Metallic taste reported during tDCS | 0 | 0 | 0
  Itching reported during tDCS | 5.6 | 2.1 | 5.7
  Pain reported during RT or OT | 5.7 | 24.3 | 7.5
  Fatigue reported during RT or OT | 18.9 | 14 | 17
  Dizziness reported during RT or OT | 0 | 0 | 0
  Syncope reported during RT or OT | 0 | 0 | 0
  Seizure reported during RT or OT | 0 | 0 | 0
  Sleepiness reported during RT or OT | 9.4 | 6.4 | 5.7
  Dysesthesia reported during RT or OT | 1.8 | 0 | 0
  Pain reported during PT | 11.3 | 23.4 | 24.5
  Fatigue reported during PT | 3.8 | 17 | 0
  Dizziness reported during PT | 0 | 0 | 0
  Syncope reported during FT | 0 | 0 | 0
  Seizure reported during PT | 0 | 0 | 0
  Sleepiness reported during PT | 1.8 | 6.4 | 5.7
  Dysesthesia reported during PT | 0 | 0 | 0

3. Secondary Outcome: Change in Modified Rankin Scale
Description: Scores range from 0 to 6. Higher scores indicate greater severity.
Time Frame: 6 weeks from baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 0 [0 to 0] | 0 [0 to -1] | -1 [-1 to -1]

4. Secondary Outcome: Change in National Institutes of Health Stroke Scale
Description: Scores range from 0 to 42. Higher scores indicate greater severity.
Time Frame: 6 weeks from baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | -3 [-5 to 0] | -1 [-2 to -1] | -2 [-3 to 0]

5. Secondary Outcome: Change in Stroke Impact Scale
Description: Scores in each domain of the Stroke Impact Scale range from 0 to 100, with higher scores indicating a better quality of life. The change was calculated as the value at the later time point minus the value at the earlier time point; so that, positive numbers represent increases and negative numbers represent decreases.
Time Frame: 6 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale
  Strength | 14.6 (7.7) | 16.7 (7.8) | 10.4 (7.7)
  Memory | 11.9 (4.4) | 14.3 (10.4) | -1.2 (3.6)
  Emotions | 9.2 (13.6) | 5.5 (3.1) | 3.7 (1.5)
  Comunication | 2.3 (6.7) | 6.0 (1.7) | 3.6 (4.4)
  Activities of daily living | 14.1 (22.4) | 25.8 (10.0) | 20.0 (7.8)
  Mobility | 24.1 (30.4) | 15.8 (1.0) | 20.4 (2.5)
  HandFunction | 15.0 (12.2) | 36.7 (0.3) | 46.6 (17.8)
  Participation | 10.4 (34.7) | 15.6 (6.6) | -6.2 (6.2)

6. Secondary Outcome: Number of Participants Who Presented Score on Modified Ashworth Scale >2
Description: Scores range from 0 to 4, with 5 choices. A score of 1 indicates no resistance, and 4 indicates rigidity.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

7. Secondary Outcome: Change in Motor Activity Log
Description: Each domain contains taks scored on 0 to 5 ordinal scale. Lower scores indicate greater severity.
Time Frame: 6 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale
  Amount of Movement | 0.6 (0.4) | 0.4 (0.4) | 0.6 (0.2)
  Quality of Movement | 0.6 (0.4) | 0.5 (0.6) | 0.8 (0.5)

8. Secondary Outcome: Upper Extremity Fugl Meyer Assessment
Description: Motor function subscale was assessed. Scores range from 0 to 66. Lower scores indicate greater severity.
Time Frame: 6 months follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 2
score on a scale | 42 (13) | 34 (14.9) | 44.5 (15.5)

9. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 6 months follow-up
Measure: Number; unit: participants
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 2
participants
  headache | 0 | 0 | 0
  pain on shoulder mobilization | 1 | 2 | 1
  dizziness | 0 | 0 | 0
  syncope | 0 | 0 | 0
  seizures | 0 | 0 | 0
  dysesthesia | 0 | 0 | 0
  psychiatric disorder | 0 | 0 | 0
  sleep | 0 | 1 | 0

10. Secondary Outcome: Change in Fatigue Severity Scale
Description: Fatigue Severity Scale is a 9 -item questionnaire. Each item scores on a 7-point scale.
  The total score range from 9 to 63 points. Higher scores indicate greater fatigue.
Time Frame: 6 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 1.7 (11.4) | -1.7 (16.3) | -30.7 (13.7)

11. Secondary Outcome: Change in Pittsburgh Sleep Quality Index
Description: The global Pittsburgh Sleep Quality Index score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21. Lower scores denote a healthier sleep quality.
Time Frame: 6 weeks from baseline
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | -1.0 (1.0) | -2.3 (2.5) | 0.3 (3.1)

ADVERSE EVENTS:
Time Frame: 06 months
Description: Data about adverse effect were collected in each session of treatment, for each different intervention - tDCS, Physical Therapy, and motor therapy (Robotic therapy or Occupational Therapy).
  All minor adverse events related (tingling, pinching, fatigue, pain, sleepiness, fatigue and pain) were considered treatment-related and reported to Ethical Committee. Two events of fall outside the hospital were related and considered non-treatment-related.
Arm/Group | Active tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Robotic Therapy + Physical Therapy | Sham tDCS + Physical Therapy + Occupational Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS + Robotic Therapy + Physical Therapy (N=3) | Sham tDCS + Robotic Therapy + Physical Therapy (N=3) | Sham tDCS + Physical Therapy + Occupational Therapy (N=3)
Tingling (Skin and subcutaneous tissue disorders) | 3 (53) | 3 (13) | 2 (20) — Tolerability to tDCS intervention
Pinching (Skin and subcutaneous tissue disorders) | 1 (5) | 3 (15) | 2 (16) — Tolerability to tDCS intervention
Fatigue (Musculoskeletal and connective tissue disorders) | 2 (10) | 2 (7) | 1 (8) — Tolerability to motor interventions (Robotic Therapy or Occupational Therapy)
Pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (11) | 2 (4) — Tolerability to motor interventions (Robotic Therapy or Occupational Therapy)
Sleepiness (Nervous system disorders) | 2 (5) | 1 (3) | 2 (3) — Tolerability to motor interventions (Robotic Therapy or Occupational Therapy)
Fatigue (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (8) | 0 (0) — Tolerability to Physical Therapy interventions
Pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (11) | 1 (13) — Tolerability to Physical Therapy interventions

LIMITATIONS AND CAVEATS:
The study was stopped earlier due to low recruitment rates. We consider psychosocial aspects and poor family support as an important factor to these low rates. The small sample size (9 patients) does not allow conclusions with statistical relevance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes